CLINICAL TRIAL: NCT01645306
Title: Revacept, an Inhibitor of Platelet Adhesion in Symptomatic Carotid Stenosis: A Phase II, Multicentre; Randomised, Dose-finding, Double-blind and Placebo Controlled Superiority Study With Parallel Groups
Brief Title: Revacept in Symptomatic Carotid Stenosis
Acronym: RevaceptCS02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AdvanceCor GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Revacept/CS/02
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Carotid Stenosis; Atherosclerosis; Stroke; Transient-ischaemic Attack; TIA; Amaurosis Fugax
MeSH Terms: conditions — Carotid Stenosis; Atherosclerosis; Stroke; Ischemic Attack, Transient; Amaurosis Fugax | interventions — Revacept; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phosphate buffered saline (PBS), 1% sucrose, 4% mannitol (Placebo Comparator): Placebo control with PBS, 1% sucrose and 4% mannitol
  Interventions: Drug: Placebo
- 40 mg Revacept (Active Comparator): low dose Revacept 40mg in PBS, 1% sucrose, 4% mannitol
  Interventions: Drug: Revacept
- 120 mg Revacept (Active Comparator): high dose revacept 120mg in PBS, 1% sucrose, 4% mannitol
  Interventions: Drug: Revacept

INTERVENTIONS:
Drug: Revacept — single intravenous injection
  Other Names: 40 mg or 120 mg
  Arms: 120 mg Revacept; 40 mg Revacept
Drug: Placebo — single intravenous injection
  Other Names: Control Group
  Arms: Phosphate buffered saline (PBS), 1% sucrose, 4% mannitol

SUMMARY:
Patients suffering from symptomatic carotid artery stenosis, transient ischemic attacks (TIAs), amaurosis fugax or stroke receive either Revacept (single dose) plus antiplatelet monotherapy or monotherapy alone.

Patients receive a single dose of trial medication by intravenous infusion for 20 minutes. Patients are followed up one and three days after treatment, at 3 months and by a telephone interview at 12 months.

DETAILED DESCRIPTION:
Patients had a more than 50% carotid artery stenosis according to ECST and suffered from ischemic stroke, transitory ischemic attack or intermittent blindness (amaurosis fugax) within the last 30 days. All patients were on standard medication with aspirin or clopidogrel and received heparin for thrombosis prophylaxis. Carotid endarterectomy (CEA), carotid stenting (CAS) or best medical therapy for treatment of the carotid stenosis and prevention of secondary thrombo-emboli was performed according to guidelines. Additional treatment with Revacept or placebo was done on top of the standard therapy. Therefore the control group receiving placebo was already on the standard medical therapy for patients with symptomatic carotid stenosis and received also the guideline conform interventions CEA, CAS or best medical therapy.

Secondary prophylaxis of thrombo-embolic ischemic events by Revacept should be investigated. Therefore microemboli were detected by transcranial Doppler and ischemic brain lesions were investigated by diffusion weighted imaging magnetic resonance imaging (DWI-MRI) scan as exploratory endpoints. Moreover clinical endpoints such as stroke, TIA, myocardial infarction, coronary intervention and death were investigated at 1 week, 3 months and 12 months follow-up. Safety was closely monitored with emphasis on bleeding complications as bleeding is the most dreaded complication of anti-thrombotic agents especially in patients with cerebral strokes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Target population

   * Diagnosis:

     * Extracranial carotid artery stenosis (diagnosed by vascular duplex ultrasound peak flow or angiography)
     * Lesions with ≥ 50 % stenosis according to the European Carotid Surgery Trial (ECST) criteria
     * TIA, amaurosis fugax or stroke within the last 30 days
   * Age and sex: Men and women aged > 18 years Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after receiving investigational product in such a manner that the risk of pregnancy is minimised.

Exclusion Criteria:

1. Sex and reproductive Status:

   * WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for up to 4 weeks after receiving investigational product.
   * Women who are pregnant or breastfeeding
   * Women with a positive pregnancy test on enrollment or prior to investigational product administration.
2. Target disease exceptions

   * NIHSS score > 18
   * Recent intracerebral haemorrhage by X-ray computed tomography (CT) or nuclear magnetic resonance (NMR)
   * Cardiac cause of embolisation (atrial fibrillation or other cardiac source e.g. artificial heart valves)
3. Medical history and concurrent disease

   * History of hypersensitivity, contraindication or serious adverse reaction to inhibitors of platelet aggregation, hypersensitivity to related drugs (cross-allergy) or to any of the excipients in the study drug
   * History or evidence of thrombocytopenia (<30.000/ul), bleeding diathesis or coagulopathy (pathological international normalised ratio (INR) or activated partial thromboplastin time (aPTT))
   * Thrombolysis within the last 48 hours
   * Relevant haemorrhagic transformation as determined by CT, NMR or anamnesis
   * Oral anticoagulation or dual anti-platelet therapy with aspirin or clopidogrel and other P2Y inhibitors at screening (3 days for dipyridamole extended release; 8 hours for tirofiban/Aggrastat)
   * Sustained hypertension (systolic BP > 179 mmHg or diastolic BP >109 mmHg)
   * History of severe systemic disease such as terminal carcinoma, renal failure (or current creatinine > 200 umol/l), cirrhosis, severe dementia, or psychosis
   * Current severe liver dysfunction (transaminase level greater than 5-fold over upper normal range limit)
   * Active autoimmune disorder such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis or glomerulonephritis
   * Known atrial fibrillation or other clinically significant ECG abnormalities (at present)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-03-08 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2019-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holger Poppert, Prof. Dr., Principal Investigator — Department of Neurology, TU Munich; Ian M Loftus, MD, Principal Investigator — St George's NHS Trust
Locations (12):
- Germany (8):
  - Site 01: Department of Neurology, TU Munich, Munich, Bavaria
  - Site 08: Universitätsklinikum Essen, Klinik für Neurologie, Essen
  - Site 11: Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Site 07: Medizinische Hochschule Hannover, Klinik für Neurologie, Hanover
  - Site 12: Universitätsklinikum Leipzig AöR, Leipzig
  - Site 09: Universitätsmedizin Mainz, Klinik und Poliklinik für Neurologie, Mainz
  - Site 04: Universitätsklinikum Tübingen, Klinik für Allgemeine Neurologie, Tübingen
  - Site 06: Universitätsklinikum Ulm, Abteilung für Neurologie, Ulm
- United Kingdom (4):
  - Site 23 - University Hospital Coventry NHS Trust, Coventry
  - Site 26 - University College London Hospital, London
  - Site 28 - King's College London Hospital, London
  - Site 20: St George's NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bultmann A, Li Z, Wagner S, Peluso M, Schonberger T, Weis C, Konrad I, Stellos K, Massberg S, Nieswandt B, Gawaz M, Ungerer M, Munch G. Impact of glycoprotein VI and platelet adhesion on atherosclerosis--a possible role of fibronectin. J Mol Cell Cardiol. 2010 Sep;49(3):532-42. doi: 10.1016/j.yjmcc.2010.04.009. Epub 2010 Apr 27. PMID 20430036
- [Background] Goertler M, Baeumer M, Kross R, Blaser T, Lutze G, Jost S, Wallesch CW. Rapid decline of cerebral microemboli of arterial origin after intravenous acetylsalicylic acid. Stroke. 1999 Jan;30(1):66-9. doi: 10.1161/01.str.30.1.66. PMID 9880390
- [Background] Markus HS, Droste DW, Kaps M, Larrue V, Lees KR, Siebler M, Ringelstein EB. Dual antiplatelet therapy with clopidogrel and aspirin in symptomatic carotid stenosis evaluated using doppler embolic signal detection: the Clopidogrel and Aspirin for Reduction of Emboli in Symptomatic Carotid Stenosis (CARESS) trial. Circulation. 2005 May 3;111(17):2233-40. doi: 10.1161/01.CIR.0000163561.90680.1C. Epub 2005 Apr 25. PMID 15851601
- [Background] Massberg S, Konrad I, Bultmann A, Schulz C, Munch G, Peluso M, Lorenz M, Schneider S, Besta F, Muller I, Hu B, Langer H, Kremmer E, Rudelius M, Heinzmann U, Ungerer M, Gawaz M. Soluble glycoprotein VI dimer inhibits platelet adhesion and aggregation to the injured vessel wall in vivo. FASEB J. 2004 Feb;18(2):397-9. doi: 10.1096/fj.03-0464fje. Epub 2003 Dec 4. PMID 14656994
- [Background] Molloy J, Markus HS. Asymptomatic embolization predicts stroke and TIA risk in patients with carotid artery stenosis. Stroke. 1999 Jul;30(7):1440-3. doi: 10.1161/01.str.30.7.1440. PMID 10390320
- [Background] Nieswandt B, Watson SP. Platelet-collagen interaction: is GPVI the central receptor? Blood. 2003 Jul 15;102(2):449-61. doi: 10.1182/blood-2002-12-3882. Epub 2003 Mar 20. PMID 12649139
- [Background] Ringelstein EB, Droste DW, Babikian VL, Evans DH, Grosset DG, Kaps M, Markus HS, Russell D, Siebler M. Consensus on microembolus detection by TCD. International Consensus Group on Microembolus Detection. Stroke. 1998 Mar;29(3):725-9. doi: 10.1161/01.str.29.3.725. PMID 9506619
- [Background] Schonberger T, Siegel-Axel D, Bussl R, Richter S, Judenhofer MS, Haubner R, Reischl G, Klingel K, Munch G, Seizer P, Pichler BJ, Gawaz M. The immunoadhesin glycoprotein VI-Fc regulates arterial remodelling after mechanical injury in ApoE-/- mice. Cardiovasc Res. 2008 Oct 1;80(1):131-7. doi: 10.1093/cvr/cvn169. Epub 2008 Jun 19. PMID 18566102
- [Background] Ungerer M, Rosport K, Bultmann A, Piechatzek R, Uhland K, Schlieper P, Gawaz M, Munch G. Novel antiplatelet drug revacept (Dimeric Glycoprotein VI-Fc) specifically and efficiently inhibited collagen-induced platelet aggregation without affecting general hemostasis in humans. Circulation. 2011 May 3;123(17):1891-9. doi: 10.1161/CIRCULATIONAHA.110.980623. Epub 2011 Apr 18. PMID 21502572
- [Background] Jamasbi J, Megens RT, Bianchini M, Munch G, Ungerer M, Faussner A, Sherman S, Walker A, Goyal P, Jung S, Brandl R, Weber C, Lorenz R, Farndale R, Elia N, Siess W. Differential Inhibition of Human Atherosclerotic Plaque-Induced Platelet Activation by Dimeric GPVI-Fc and Anti-GPVI Antibodies: Functional and Imaging Studies. J Am Coll Cardiol. 2015 Jun 9;65(22):2404-15. doi: 10.1016/j.jacc.2015.03.573. PMID 26046734
- [Background] Kleiman NS, Kolandaivelu K. Expanding the Roster: Developing New Inhibitors of Intravascular Thrombosis. J Am Coll Cardiol. 2015 Jun 9;65(22):2416-9. doi: 10.1016/j.jacc.2015.03.576. No abstract available. PMID 26046735
- [Derived] Uphaus T, Richards T, Weimar C, Neugebauer H, Poli S, Weissenborn K, Imray C, Michalski D, Rashid H, Loftus I, Rummey C, Ritter M, Hauser TK, Munch G, Groschel K, Poppert H. Revacept, an Inhibitor of Platelet Adhesion in Symptomatic Carotid Stenosis: A Multicenter Randomized Phase II Trial. Stroke. 2022 Sep;53(9):2718-2729. doi: 10.1161/STROKEAHA.121.037006. Epub 2022 Jun 13. PMID 35695006

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Phosphate buffered saline (PBS), 1% sucrose, 4% mannitol
  Placebo: single intravenous injection
- 40 mg Revacept: 40 mg Revacept in phosphate buffered saline (PBS), 1% sucrose, 4% mannitol
  Revacept: single intravenous injection
- 120 mg Revacept: 120 mg in phosphate buffered saline (PBS), 1% sucrose, 4% mannitol
  Revacept: single intravenous injection
Period: Overall Study
Arm/Group | Placebo | 40 mg Revacept | 120 mg Revacept
Started | 51 | 54 | 53
Completed | 49 | 50 | 48
Not Completed | 2 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- 120 mg Revacept: 120 mg Revacept in phosphate buffered saline (PBS), 1% sucrose, 4% mannitol
  Revacept: single intravenous injection
- Total: Total of all reporting groups
Arm/Group | Placebo | 40 mg Revacept | 120 mg Revacept | Total
Number analyzed (Participants) | 51 | 54 | 53 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (10.25) | 68.7 (10.45) | 68.4 (9.82) | 68.1 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 17 | 38
  Male | 43 | 41 | 36 | 120
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Origin: African | 1 | 0 | 0 | 1
  Ethnic Origin: Asian | 1 | 2 | 0 | 3
  Ethnic Origin: Caucasian | 49 | 52 | 53 | 154
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14 | 18 | 18 | 50
  Germany | 37 | 36 | 35 | 108

OUTCOME MEASURES:

1. Primary Outcome: New DWI Lesion(s)
Description: The number of new diffusion weighted imaging (DWI) lesion(s) reported. (1 day after intervention compared to baseline).
Time Frame: 1 day post intervention
Measure: Mean (Standard Deviation); unit: Number of new lesions
Groups:
- 40 mg Revacept; 120 mg Revacept: in phosphate buffered saline (PBS), 1% sucrose, 4% mannitol
  Revacept: single intravenous injection
Arm/Group | Placebo | 40 mg Revacept | 120 mg Revacept
Number analyzed (Participants) | 51 | 54 | 53
Number of new lesions | 1.2 (0.4) | 1.0 (0.3) | 0.6 (0.3)

2. Other Pre Specified Outcome: Patients With Any Stroke or Transient Ischemic Attack (TIA)
Description: patients with any stroke or TIA occuring within 90 days after IMP application.
Time Frame: 90 days after IMP application
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Revacept | 120 mg Revacept
Number analyzed (Participants) | 51 | 54 | 53
Participants | 6 | 6 | 4

3. Other Pre Specified Outcome: Major Bleedings
Description: patients with major bleedings occuring within 90 days after IMP application
Time Frame: 90 days after IMP application
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Revacept | 120 mg Revacept
Number analyzed (Participants) | 51 | 54 | 53
Participants | 5 | 6 | 4

4. Other Pre Specified Outcome: Any Clinical Event
Description: patients with any stroke & TIA, myocardial infarction & percutaneous coronary intervention (PCI), death or bleeding within one year (365 days) after IMP application.
Time Frame: 365 days after IMP application
Measure: Number; unit: Number of Events
Arm/Group | Placebo | 40 mg Revacept | 120 mg Revacept
Number analyzed (Participants) | 51 | 54 | 53
Number of Events | 19 | 15 | 10

5. Other Pre Specified Outcome: Anti-Drug Antibodies
Description: Anti-drug antibodies were measured at baseline and 3 month after IMP application.
  Number of patients with positive anti-drug antibodies compared to baseline are counted.
Time Frame: 3 month (+/- 1 month) after IMP application
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 40 mg Revacept | 120 mg Revacept
Number analyzed (Participants) | 51 | 54 | 53
Participants | 0 | 0 | 0

6. Other Pre Specified Outcome: Participants With Adverse Events (AEs)
Description: All adverse events were assessed during complete study period (~ 1 year after IMP application).
Time Frame: ~ 365 days after IMP application (whole study period)
Measure: Number; unit: participants
Arm/Group | Placebo | 40 mg Revacept | 120 mg Revacept
Number analyzed (Participants) | 51 | 54 | 53
participants
  patients with adverse events | 35 | 41 | 32
  patients with drug related AEs | 4 | 10 | 2
  patients with serious AEs | 17 | 17 | 15
  patients with drug related serious AEs | 1 | 4 | 0
  patients with AE with fatal outcome events | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse Event Data was gathered at a 3 month follow up visit in the clinic and up to one year by a telephone interview.
Arm/Group | Placebo | 40 mg Revacept | 120 mg Revacept
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/54 | 1/53
Serious Adverse Events (participants affected / at risk) | 17/51 | 17/54 | 15/53
Other Adverse Events (participants affected / at risk) | 18/51 | 24/54 | 17/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | 40 mg Revacept (N=54) | 120 mg Revacept (N=53)
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0
Ischemia (Vascular disorders) | 0 | 0 | 1
Carotid Endarterectomy (Surgical and medical procedures) | 0 | 1 | 1
Chemotherapy (Surgical and medical procedures) | 1 | 0 | 0
Coronary angioplasty (Surgical and medical procedures) | 0 | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1 | 0
Skin lesion removal (Surgical and medical procedures) | 0 | 1 | 0
Vocal cordectomy (Surgical and medical procedures) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Sarcoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Cerebral hyperperfusion syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Angiocardiogram (Investigations) | 0 | 1 | 0
Biopsy larynx (Investigations) | 0 | 1 | 0
Cardiac clearance (Investigations) | 1 | 0 | 0
Diffusion-weighted brain MRI (Investigations) | 0 | 0 | 1
Weight decrease (Investigations) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 2 | 2
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 2 | 1
Cerebral ischemia (Nervous system disorders) | 2 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Clumsiness (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Parkinsonism (Nervous system disorders) | 1 | 0 | 0
Postictal paralysis (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1 | 0
Stroke in evolution (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 1 | 4
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc prorusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | 40 mg Revacept (N=54) | 120 mg Revacept (N=53)
Hypertension (Vascular disorders) | 4 | 2 | 2
Oedama peripheral (General disorders) | 2 | 5 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 3 | 1 | 2
Cardiac murmur (Investigations) | 3 | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 3
Transient ischaemic attack (Nervous system disorders) | 2 | 1 | 4
Nausea (Gastrointestinal disorders) | 1 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Pneumonia (Infections and infestations) | 4 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 2

LIMITATIONS AND CAVEATS:
The study was originally planned as primary endpoint study for the evaluation of reduction of micro-embolic signals (MES) by transcranial Doppler (TCD). Therefore MES incidence was a key inclusion criteria at screening. Due to low incidence of MES in this patient population with high screening failure rate the mandatory presence of MES was abandoned during the course of the study. Consecutively the study was changed to an explorative study of the same protocol specified endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-06-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT01645306/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT01645306/SAP_001.pdf